CLINICAL TRIAL: NCT01005576
Title: A Pilot Trial of Unrelated Donor Hematopoietic Cell Transplantation for Children With Severe Thalassemia Using a Reduced Intensity Conditioning Regimen (The URTH Trial)
Brief Title: Reduced Intensity Transplant Conditioning Regimen for Severe Thalassemia
Acronym: URTH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Carelon Research (Other); Pediatric Blood and Marrow Transplant Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCRN-NMD 0901
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Severe Thalassemia
Keywords: Thalassemia; Alemtuzumab; Hematopoietic cell transplant; non-myeloablative
MeSH Terms: conditions — Thalassemia | interventions — fludarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conditioning regimen (Experimental): Hydroxyurea days -50 to -21 Alemtuzumab days -21 to -19 Fludarabine days -8 to -4 Thiotepa day -4 Melphalan day -3 Stem cell infusion day 0
  Interventions: Drug: Transplant conditioning regimen of alemtuzumab, fludarabine, and melphalan

INTERVENTIONS:
Drug: Transplant conditioning regimen of alemtuzumab, fludarabine, and melphalan — Days -50 to -21: Hydroxyurea 30mg/kg po Day -22: Alemtuzumab 3mg IV Day -21: Alemtuzumab 10mg IV Day -20: Alemtuzumab 15mg IV Day -19: Alemtuzumab 20mg IV Day -8: Fludarabine 30mg/m2 IV Day -7: Fludarabine 30mg/m2 IV Day -6: Fludarabine 30mg/m2 IV Day -5: Fludarabine 30mg/m2 IV Day -4: Fludarabine 30mg/m2 IV Day -4: Thiotepa 8mg/kg IV Day -3: Melphalan 140mg/m2 IV Day 0: Stem cell infusion

SUMMARY:
This study is being done to determine if blood cell transplants, with either bone marrow or cord blood from unrelated donors, are effective in children with severe thalassemia and if this treatment approach has acceptable risks and side effects.

This study includes a preparative regimen with Hydroxyurea, Alemtuzumab, Fludarabine, Thiotepa and Melphalan that provides intense host immunosuppression without myeloablation. The primary hypothesis is that this regimen will promote stable engraftment of unrelated donor hematopoietic cells, support normal erythropoiesis, and result in an event free survival of > 75% of children with thalassemia major.

ELIGIBILITY:
Inclusion Criteria:

* 1-16.00 years old
* Have transfusion dependent thalassemia major
* Shall not have an HLA-matched family donor
* Must have a suitably matched unrelated marrow donor or UCB product
* Lansky score >/= 70
* Adequate pulmonary, renal, liver, and other organ function as defined in protocol
* Negative pregnancy test
* Adequate total nucleated cell or CD34+ dose of product as defined in protocol
* Iron chelation must be discontinued >/= 48 hours prior to conditioning regimen

Exclusion Criteria:

* Pregnant or breastfeeding
* HIV positive
* Prior allogeneic marrow or stem cell transplantation

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Shenoy, MD, Principal Investigator — Washington University School of Medicine
Locations (18):
- United States (18):
  - Regents of University of California- UCLA, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - All Children's Research Institute, Inc., St. Petersburg, Florida
  - Emory University, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 11 academic medical centers. The first participant was enrolled in May 2010 and the last participant was enrolled in April 2012.
Period: Overall Study
Arm/Group | Conditioning Regimen
Started | 21
Completed | 21 (All participants completed the conditioning regimen and received their stem cell transplant)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Conditioning Regimen
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 10 [1.8 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 5
  Race/Ethnicity: Middle Eastern | 2
  Race/Ethnicity: African American | 1
  Race/Ethnicity: Hispanic | 2
  Race/Ethnicity: Pakistani | 2
  Race/Ethnicity: Caucasian | 3
  Race/Ethnicity: Vietnamese | 1
  Race/Ethnicity: More than 1 race reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Primary Objective: Event-free Survival at 1 Year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Regimen
Number analyzed (Participants) | 21
Participants | 17

2. Secondary Outcome: Development of Graft Versus Host Disease (GVHD)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Regimen
Number analyzed (Participants) | 21
Participants
  Participants who developed any GVHD | 12
  Participants who did not develop any GVHD | 9

3. Secondary Outcome: Median Time to ANC Engraftment
Time Frame: 100 days
Measure: Median (Full Range); unit: days
Arm/Group | Conditioning Regimen
Number analyzed (Participants) | 21
days | 14 [10 to 46]

4. Secondary Outcome: Median Time to Platelet Engraftment
Time Frame: 100 days
Population: 3 participants did not engraft platelets
Measure: Median (Full Range); unit: days
Arm/Group | Conditioning Regimen
Number analyzed (Participants) | 18
days | 27.5 [18 to 234]

5. Secondary Outcome: Incidence of Disease Recurrence
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Conditioning Regimen
Number analyzed (Participants) | 21
Participants | 1

ADVERSE EVENTS:
Arm/Group | Conditioning Regimen
All-Cause Mortality (participants affected / at risk) | 4/21
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning Regimen (N=21)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 4 — Respiratory distress, pulmonary failure, pulmonary hemorrhage
Pain (General disorders) | 1
Graft rejection (General disorders) | 1
Edema (General disorders) | 1 — Head and neck edema
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning Regimen (N=21)
CMV reactivation (Infections and infestations) | 14
Veno Occlusive Disease (Hepatobiliary disorders) | 1
Hyperbilirubinemia (Investigations) | 1
Hypercalcemia (Investigations) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Infection (other than CMV) (Infections and infestations) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No